CLINICAL TRIAL: NCT07341451
Title: Novel Experimental Methods to Measure Apically Extruded Debris and Solutions During Root Canal Intstrumantation, an Invitro Study
Brief Title: Measuring Apical Debris Extrusion With a Novel Laboratory Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Selenay Ucas Yildiz (Other)
Collaborators: necmettin erbakan university Scientific Research Projects (BAP) (Unknown)
Responsible Party: Sponsor-Investigator, Fatma Selenay Ucas Yildiz, Research Assistant and Principal Investigator, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025/539; 23068 (Other: Necmettin Erbakan University, Faculty of Dentistry, Clinical Sciences Ethics Committee)
Record Dates: First submitted 2025-10-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Apical Extrusion During Root Canal Treatment
Keywords: Debris extrusion; Irrigant extrusion; ProTaper Next; ProTaper Gold; Apical extrusion; Chromium-cobalt particles; Metal particles; Barium sulfate; Radiopacity

STUDY DESIGN:
Intervention Model Description: Eighty extracted human mandibular premolars were randomly assigned into four parallel groups (n=20 each) to evaluate apical extrusion of debris and irrigants using two different rotary systems (ProTaper Gold, ProTaper Next) and two evaluation methods (metal particles for debris, barium sulfate solution for irrigants)
Who Masked: Outcomes Assessor
Masking Description: During root canal instrumentation, the operator could not observe the amount of extruded debris or irrigant. Radiographic evaluation of extrusion was performed afterwards. Although the assessor was aware of group allocation, the extrusion itself was not visible during instrumentation, thus minimizing bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ProTaper Gold - Debris Extrusion (Experimental): Extracted mandibular premolars shaped with ProTaper Gold rotary files.
  Apical extrusion of debris measured using chromium-cobalt particles.
  Interventions: Device: ProTaper Gold Rotary File System
- ProTaper Next - Debris Extrusion (Experimental): Extracted mandibular premolars shaped with ProTaper Next rotary files.
  Apical extrusion of debris measured using chromium-cobalt particles.
  Interventions: Device: ProTaper Next Rotary File System
- ProTaper Gold - Irrigant Extrusion (Experimental): Extracted mandibular premolars shaped with ProTaper Gold rotary files.
  Apical extrusion of irrigant measured using barium sulfate-enhanced NaOCl.
  Interventions: Device: ProTaper Gold Rotary File System
- ProTaper Next - Irrigant Extrusion (Experimental): Extracted mandibular premolars shaped with ProTaper Next rotary files.
  Apical extrusion of irrigant measured using barium sulfate-enhanced NaOCl
  Interventions: Device: ProTaper Next Rotary File System

INTERVENTIONS:
Device: ProTaper Gold Rotary File System — Root canal instrumentation performed using ProTaper Gold rotary file system at working length. Files were used in sequence (S1, F1-F3) following the manufacturer's instructions for torque and rpm. Irrigation was performed with NaOCl during shaping
  Arms: ProTaper Gold - Debris Extrusion; ProTaper Gold - Irrigant Extrusion
Device: ProTaper Next Rotary File System — Root canal instrumentation performed using ProTaper Next rotary file system at working length. Files were used in sequence (X1-X3) following the manufacturer's instructions for torque and rpm. Irrigation was performed with NaOCl during shaping
  Arms: ProTaper Next - Debris Extrusion; ProTaper Next - Irrigant Extrusion

SUMMARY:
Endodontic treatment occupies a critical role in dentistry, serving to prolong the longevity of teeth within the oral cavity and prevent early tooth loss. This treatment is particularly indicated in cases where the pulp tissue is infected or has suffered damage. The primary objective of endodontic treatment is to clean the infected pulp tissue, shape the root canals, and adequately fill these spaces to preserve the functionality of the tooth. A successful endodontic procedure is essential not only for ensuring the longevity of the tooth but also for delaying resorption in surrounding tissues. Furthermore, it allows the patient to maintain masticatory function without losing proprioceptive sensation, which is a key indicator of the treatment's success.

During root canal instrumentation, there is a risk of necrotic debris, microorganisms, and dentin particles being displaced through the apical foramen into the periapical tissue. This displacement can increase the risk of infection and lead to postoperative complications. The preservation of the apical foramen is one of the most critical stages in the endodontic treatment process. Materials that extrude beyond the apical foramen can cause irritation and inflammation in the alveolar bone. This situation may exacerbate postoperative pain and discomfort, negatively affecting the patient's satisfaction with the treatment. Additionally, such displacements can compromise the overall success of the procedure by increasing the risk of reinfection. Therefore, preventing these displacements during root canal shaping is a factor that directly influences the success of the treatment.

In the literature, precision scales are commonly used to measure the materials displaced from the apex. However, there are discrepancies regarding the reliability of these scales, particularly concerning their measurement accuracy for very small quantities. It has been observed that these precision scales may not provide sufficient accuracy in certain situations, making it challenging to accurately determine the amount of extruded materials. This issue poses a significant barrier to the assessment of endodontic treatment outcomes. Consequently, there is a need for the development of existing measurement methods and the exploration of alternative approaches. The integration of new technologies for measuring the quantity of extruded materials could enhance the understanding and management of treatment processes.

In this context, the primary aim of this research is to develop new methods for the more accurate and reliable measurement of materials displaced from the apex. Novel measurement techniques will allow for a more precise determination of the quantity of extruded materials, thereby enhancing the efficacy of endodontic treatment processes. Furthermore, this research aims to contribute to the reduction of postoperative complications and improve patient satisfaction during the treatment process. Ultimately, innovative approaches of this nature are of great importance for the success of endodontic treatments and patient satisfaction. Research in the field of endodontics will not only guide clinical practices but also make significant contributions to the scientific literature. Such innovations will assist in the development of future treatment protocols and the enhancement of patient care.

DETAILED DESCRIPTION:
Detailed Description

The purpose of this study is to develop alternative and reliable measurement methods for quantifying solid and liquid substances unintentionally extruded from the apical foramen during endodontic treatment with higher precision. The investigators will assess the limitations and applicability of the proposed methods, which are expected to contribute to future treatment improvements. The study also aims to evaluate the potential of these methods to reduce postoperative pain and infection risks in clinical practice. This research is anticipated to make significant contributions to enhancing the effectiveness and reliability of endodontic treatment processes.

This in vitro study was designed to evaluate the amount of apical extrusion (debris and irrigation solution overflow) occurring during root canal treatment. A total of 80 extracted human lower premolar teeth, selected according to predefined criteria, were used. The primary objective was to compare the effects of two different rotary file systems-ProTaper Gold and ProTaper Next-on the amount of apical overflow.

Selection and Preparation of Specimens

The specimens consisted of extracted lower premolars with fully developed roots, a single canal, a single apical foramen, moderate root inclination, and no previous endodontic treatment. Root canal inclination angles were determined using the Schneider method, and only specimens with inclinations between 5° and 20° were included to better simulate clinical conditions. Teeth with multiple apical foramina, cracks, or fractures were excluded following examination under magnification. The criteria of single root and single canal were verified radiographically.

Disinfection and Preparation

Teeth were disinfected in 5% sodium hypochlorite for 10 minutes, rinsed with distilled water, and stored in physiological saline. Standard endodontic access cavities were prepared, and canal orifices were identified using an endodontic explorer. Pulp remnants were removed with hand files. The working length was standardized to 0.5 mm short of the anatomical apex for all specimens.

Root Canal Preparation and Standardization

Initial shaping was performed with a ProTaper Gold S1 file using the manufacturer's recommended speed and torque settings. Irrigation with 2 ml sodium hypochlorite was applied during instrumentation. Specimens in which a #20 K-file could pass through the apical foramen were excluded to maintain standardization.

Chromium-cobalt particles were compacted into the canals to assess the apical extrusion of debris radiographically. The particles were inserted using an excavator and pluggers, ensuring homogeneous distribution. After radiographic confirmation, each specimen was placed into the experimental setup.

Experimental Setup

Each tooth was mounted on an acrylic block with its apical region in contact with a moisture-absorbing sponge that simulated periodontal tissues. This setup provided a radiolucent background for the radiographic detection of extruded materials and allowed fluid absorption, enabling blinded assessment.

Groups and Experimental Procedure

Eighty specimens were randomly assigned into four groups (n = 20) as follows:

Group 1: Debris overflow - ProTaper Gold

Group 2: Debris overflow - ProTaper Next

Group 3: Solution overflow - ProTaper Gold

Group 4: Solution overflow - ProTaper Next

Access cavities and pulp chambers were left unsealed to reflect clinical conditions.

Debris Overflow Groups (Groups 1 and 2) Root canals were instrumented to working length using ProTaper Gold or ProTaper Next files. Irrigation with 2 ml NaOCl was performed at each file stage, followed by a final rinse with 6 ml NaOCl for 3 minutes. Extruded particles were visualized radiographically and quantified using ImageJ software.

Solution Overflow Groups (Groups 3 and 4) To opacify irrigation solutions, barium sulfate powder was added to NaOCl and EDTA. The canals were instrumented with ProTaper Gold or ProTaper Next systems using these opacified irrigants. The amount of extruded solution was recorded radiographically and analyzed in ImageJ.

Data Collection and Analysis

Digital radiographs of all samples were obtained at a standardized 15 cm distance. The radiographs were evaluated blindly, and the surface area and density of extruded opaque materials were measured as percentages. Data were recorded in Excel spreadsheets and prepared for statistical analysis.

Contribution of the Study

This study introduces a novel radiographic approach for assessing apical extrusion. The use of chromium-cobalt particles and barium sulfate-enhanced irrigants enables objective visualization of extruded material, while the moisture-absorbing sponge system effectively simulates periodontal conditions. The findings are expected to facilitate the comparison of rotary file systems in terms of apical extrusion and to support the development of more reliable and clinically applicable endodontic procedures.

ELIGIBILITY:
Inclusion Criteria:

Extracted human mandibular premolars with fully formed apices Single straight root canal confirmed radiographically No resorption, fracture, or previous endodontic treatment No caries or restorations extending into the root canal

Exclusion Criteria:

Teeth with multiple canals, severe curvature (>20°) Immature apices or open apex External or internal root resorption Presence of root fractures, cracks, or structural anomalies Teeth with previous endodontic instrumentation or obturation Teeth with extensive coronal defects that compromise standardization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Radiographic Area of Apically Extruded Debris | Baseline
  During the single experimental session of root canal instrumentation and irrigation
Radiographic Area of Apically Extruded Irrigant | Baseline
  Quantification of apically extruded irrigant using barium sulfate-enhanced NaOCl/EDTA solutions. After instrumentation, standardized digital radiographs are analyzed in ImageJ to measure the radiopaque area and spread pattern of the extruded irrigant on the sponge background.

CONTACTS AND LOCATIONS:
Overall Officials: Arslan Terlemez, DDS, PhD, Study Director — Necmettin Erbakan University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Necmettin Erbakan University Faculty of Dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not involve human participants or individual participant data. All experiments were performed on extracted teeth in a laboratory setting. Therefore, no IPD will be generated or shared.

REFERENCES:
- See also: Related Info — https://erbakan.edu.tr/tr/birim/dis-hekimligi-fakultesi